CLINICAL TRIAL: NCT02831452
Title: Relationship Among Vaginal Palpation, Vaginal Squeeze Pressure and Dynamometry of Nulliparous Pelvic Floor Muscles
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Paula Magalhães Resende, PhD, Federal University of Uberlandia
Other Study IDs: 1061162/2014 CEP/UFU
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Correlation of Pelvic Floor Muscle Evaluation Methods
Keywords: pelvic floor muscles; evaluation; dynamometer; perineometer

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (4):
- non-pregnant nulliparous: nulliparous without previous gestation. Pelvic floor muscle evaluation by means of vaginal palpation, vaginal squeeze pressure (perineometer), and pelvic floor muscle strength using a proper vaginal dynamometer.
  Interventions: Other: pelvic floor muscle strength evaluation
- primigravid on 1º trimester: nulliparous women on her first pregnancy and gestational age until 13 weeks and 6 days.
  Pelvic floor muscle evaluation by means of vaginal palpation, vaginal squeeze pressure (perineometer), and pelvic floor muscle strength using a proper vaginal dynamometer.
  Interventions: Other: pelvic floor muscle strength evaluation
- primigravid on 2º trimester: nulliparous women on her first pregnancy and gestational age between 14 weeks and 27 weeks.
  Pelvic floor muscle evaluation by means of vaginal palpation, vaginal squeeze pressure (perineometer), and pelvic floor muscle strength using a proper vaginal dynamometer.
  Interventions: Other: pelvic floor muscle strength evaluation
- primigravid on 3º trimester: nulliparous women on her first pregnancy and gestational age above 28 weeks. Pelvic floor muscle evaluation by means of vaginal palpation, vaginal squeeze pressure (perineometer), and pelvic floor muscle strength using a proper vaginal dynamometer.
  Interventions: Other: pelvic floor muscle strength evaluation

INTERVENTIONS:
Other: pelvic floor muscle strength evaluation

SUMMARY:
The aim of this study is to determine if there is a correlation between digital palpation, perineometry and dynamometry as PFM function evaluation methods in nulliparous without pelvic floor dysfunction.

DETAILED DESCRIPTION:
Study design - this study was conducted in Cinesiofunctional Performance Laboratory Pelvic and Women's Health at the Federal University of Uberlandia (UFU), the volunteers were recruited from December 2014 to July 2015. This is an observational, cross-sectional and comparative study, the sample consisted of 141 nulliparous women (non-pregnant nulliparous or primigravids). All volunteer shave signed an informed consent and the study was approved by the Ethics Committee of the Federal University of Uberlandia (No.1067162/2014). Female students of UFU were invited by personal contact to participate in the study. The primigravids were participants in the Prenatal Program of the public health system in Uberlandia city and they have also been invited by personal contact. Inclusion criterion for volunteers were: never have passed for childbirth situation,ability to contract correctly the PFM and without urogynecological complaints. Exclusion criterion were: history of previous pelvic surgery, without previous sexual intercourse, and present neuromuscular diseases. The experient examiner, with expertise in PFM evaluation conducted the evaluations. After checking that they were eligible to participate in the survey, participants were asked to empty the bladder and to remain in the supine position on an appropriate bed with hips and knees flexed and maintaining the lumbar spine in neutral position.The PFM assessment was performed by vaginal palpation, vaginal squeeze pressure and dynamometry. The vaginal palpation and vaginal squeeze pressure are widely used in research involving the female pelvic floor and many studies have shown its reproducibility and validity(10, 11, 12, 13). The measurements performed with a dynamometer in this study were similar to the study of Martinho et al(4) which used the same instrument and have demonstrated reproducibility of the assessment method. During all PFM assessments, the volunteer was advised to stay relaxed and breathing normally. To be considered valid, the cranial elevation movement was observed by the examiner, as well as the absence of visible contractions of the adductor, muscles of the hip, gluteal muscles or abdominals. Strong verbal command was adopted to request the PFM contraction in all exams.

Assessments began after explaining how to perform the PFM contraction. The vaginal palpation was always the first exam to check the PFM contraction ability and then the order of vaginal squeeze pressure exam and dynamometry was randomized.

The PFM assessment by digital palpation was performed as proposed by Laycock and Jerwood. The physiotherapist introduced the index and middle fingers about 4 cm inside the vagina, and requested to hold the maximum contraction of the PFM, according to the instruction of a movement "inward and up" with the greatest possible strength. Muscle function was classified by the Oxford Scale Modified, which varies from zero (absence of muscle contraction) to five (strong contraction). The vaginal squeeze pressure was measured through Peritron equipment (Cardio Design Pty Ltd, Oakleigh, Victoria, Australia) equipped with a vaginal probe that has been covered with a non-lubricated condom and then the probe was lubricated with hypoallergenic gel. The probe sensor was connected to a microprocessor hand with a latex tube, which allows the measurement of nip pressure in centimeters of water (cmH2O). To obtain the measurements, the subjects remained positioning and vaginal sensor was introduced approximately 3.5cm into the vaginal cavity. Then the device was inflated to 100cmH2O (calibration). The female volunteers were oriented and motivated verbally to perform three voluntary maximal contractions sustained for five seconds and one minute interval between them. The correct contraction was checked visually by the physiotherapist. All volunteers were instructed to avoid using the abdominal muscles, gluteal and hip adductor. For statistical analysis, the investigator used the peak pressure provided by the equipment. The PFM contraction strength was assessed by vaginal dynamometer EMG System do Brasil (model DFV 020.101/10). It is cylindrical in shape (9.5 cm in length and 3.3 cm in diameter), made of steel and is equipped with a load cell 2 cm from its base, which can measure anteroposterior unidirectional compressive strength in Kg/force (Kgf). The equipment was previously coated with a condom and lubricated with hypoallergenic gel, which was inserted into the vaginal cavity with the load cell positioned so that it could capture the anteroposterior compression strength. The participant was asked to perform three maximal voluntary PFM contractions for eight seconds with a rest period of 30 seconds between the contractions. The same precautions for correct contraction were adopted. The best value of maximum strength (difference between the highest and lowest strength in Kgf) was used for statistical analysis. Statistical analysis was performed using Statistical Package for Social Sciences software (SPSSV17, Chicago, IL). Data normality was tested by the Shapiro-Wilk test.

To verify the correlation between the variables, the Pearson correlation test was used. Values of p < 0.05 were considered significant. The correlation values were interpreted according to the following guidelines: 0.00 - 0.19= no to slight; 0.20-0.39= mild; 0.40-0.69= moderate; 0.70-0.89= high and 0.90-1.00= very high. Data were expressed as mean and standard deviation (SD).

ELIGIBILITY:
Inclusion Criteria:

* never have passed for childbirth situation
* ability to contract correctly the PFM
* without urogynecological complaints

Exclusion Criteria:

* history of previous pelvic surgery
* without previous sexual intercourse
* present neuromuscular diseases

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: healthy women without previous labor and delivery - non-pregnant or in their first pregnancy
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
correlation between pelvic floor muscle strength evaluation methods | seven months

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Uberlândia, Uberlândia, Minas Gerais, Brazil